CLINICAL TRIAL: NCT06818916
Title: Efficacy and Safety of Hetrombopag in Promoting Platelet Engraftment After Autologous Hematopoietic Stem Cell Transplantation in Children With Neuroblastoma
Brief Title: Hetrombopag in Promoting Platelet Engraftment After Auto-HSCT in Children With Neuroblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Jun Yang, Beijing Children's Hospital, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: [2024]-Y-002-D
Record Dates: First submitted 2024-06-20; First posted 2025-02-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Delayed Platelet Engraftment; Neuroblastoma; Autologous Hematopoietic Stem Cell Transplantation
Keywords: Hetrombopag; delayed platelet engraftment; neuroblastoma; pediatrics; autologous hematopoietic stem cell transplantation
MeSH Terms: conditions — Neuroblastoma | interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — Patients enrolled were administered Hetrombopag starting from +4d after transplantation on routine medication of recombinant human thrombopoietin injection (rhTPO). The starting dose of Hetrombopag is 2.5mg or 5mg, oral, once daily (starting at 5mg/d for body weight>20kg; starting from 2.5mg/d for body weight ≤ 20kg). Adjust the dosage based on platelet count every two weeks, with a maximum dose of 7.5mg per day. Stop the medication after 6 weeks of continuous use or when PLT reaches 100 × 10^9/L.

SUMMARY:
The goal of this clinical trial is to learn if hetrombopag promotes platelet engraftment in neuroblastoma children undergoing autologous hematopoietic stem cell transplantation. The main question it aims to answer is:

· Does drug hetrombopag promote platelet engraftment? Participants will take hetrombopag every day for 6 weeks or until platelet > 100*10^9/L.

ELIGIBILITY:
Inclusion Criteria:

* Age<18 years old;
* Diagnosed as neuroblastoma;
* ECOG ≤ 2;
* First time receiving autologous hematopoietic stem cell transplantation;
* The subjects or their legal guardians agree to participate and sign the informed consent form.

Exclusion Criteria:

* ALT/AST > 3 ULN, or TBIL > 1.5 ULN;
* Have experienced congestive heart failure, arrhythmia, peripheral arteriovenous thrombosis requiring medication treatment within one year prior to enrollment, or have experienced myocardial infarction or cerebral infarction within three months prior to enrollment;
* Suffering from thromboembolic diseases;
* Other situations that are not suitable for inclusion in the study determined by researchers.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Accumulated platelet engraftment rate | From enrollment to 60 days post-transplant
  Platelet engraftment is defined as a continuous 7-day PLT ≥ 20 × 10^9/L without platelet infusion.

SECONDARY OUTCOMES:
Number of platelet transfusions | From enrollment to 60 days post-transplant
Time to platelet engraftment | From enrollment to 60 days post-transplant
progression-free survival (PFS) | From enrollment to 60 days post-transplant
  The time from enrollment to the first occurrence of disease progression or death from any cause
Adverse events | From medication to 30 days after discontinuation
  Any adverse events within 30 days of discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Stem Cell Transplantation, Beijing Children's Hospital, Capital Medical University, Beijing, China